CLINICAL TRIAL: NCT05014204
Title: Safety and Feasibility of Endoscopic Application of a Novel Therapy for Duodenal Mucosal Regeneration in the Treatment of Type II Diabetes
Brief Title: Safety and Feasibility of Novel Therapy for Duodenal Mucosal Regeneration for Type II Diabetes
Acronym: REGENT-1-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endogenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 346
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Diabetes; Diabetes Type 2; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Diabetes Mellitus
Keywords: Endoscopy; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Interventional (Experimental): All eligible patients will receive the endoscopic Endogenex procedure.
  Interventions: Device: The Endogenex Device

INTERVENTIONS:
Device: The Endogenex Device — The Endogenex device is designed to induce duodenal mucosal regeneration using pulsed electric field. The Endogenex procedure is a non-surgical, endoscopic procedure.

SUMMARY:
This is a multi-center, open-label study to assess the feasibility and preliminary safety of the Endogenex Device for endoscopic duodenal mucosal regeneration in patients with type 2 Diabetes inadequately controlled on 2-3 non-insulin glucose-lowering medications.

DETAILED DESCRIPTION:
Individuals who sign the informed consent will be screened for study eligibility. Eligible participants will be treated with the Endogenex procedure and followed up for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 22- 65 years of age
2. Current diagnosis of T2D
3. History of T2D for at least 3 years and less than or equal to 10 years
4. HbA1C of 7.5-10.0%, inclusive
5. BMI 24-40 kg/m2, inclusive
6. On two to three non-insulin glucose lowering mediations, with one at maximum tolerated dose and another at half-maximum dose at least, with no changes in medication for at least 12 weeks prior to baseline visit prior to baseline visit
7. History of failed attempt to reach glycemic goal by lifestyle modifications
8. Weight stability (defined as a < 5% change in body weight) for at least 12 weeks prior to the screening visit
9. Agree not to donate blood during participation in the study.
10. Able to comply with study requirements and understand and sign the Informed Consent Form
11. Women of childbearing potential must be using an acceptable method of contraception throughout the study
12. Willing and able to use CGM for the duration of the study and comply with study visits and study tasks as required per protocol.
13. Proof of COVID 19 vaccination.

Exclusion Criteria:

1. Diagnosed with type 1 diabetes
2. History of diabetic ketoacidosis or hyperosmolar nonketotic coma
3. Probable insulin production failure, defined as overnight fasting C-peptide serum <1 ng/mL (333pmol/l).
4. Previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes) in last 2 years.
5. Current use of insulin
6. Hypoglycemia unawareness
7. History of ≥1 severe hypoglycemia episode (defined by needing for third-party assistance) in past 6 months from the screening visit
8. Known autoimmune disease, as evidenced by a positive anti-glutamic acid decarboxylase (GAD) test, including but not limited to celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder. (Participants with adequately controlled primary hypothyroidism may be included).
9. Previous GI surgery that has changed GI anatomy or could limit treatment of the duodenum, such as Billroth 2, Roux-en-Y gastric bypass, gastric band or other similar procedures or conditions.
10. Known history of a structural or functional disorder of the upper GI tract that may impede passage of the device through the upper GI tract or increase risk of tissue damage during an endoscopic procedure, including esophagitis, stricture/stenosis, varices, diverticula, or other disorder of the esophagus, stomach and duodenum.
11. Active H. pylori infection (Participants with active H. pylori may continue with the screening process if they are treated with an appropriate antibiotic regimen)
12. History of, or gastrointestinal symptoms suggestive of gastroparesis.
13. Acute gastrointestinal illness in the previous 7 days
14. Known history of irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease and Celiac disease
15. History of chronic or acute pancreatitis.
16. Known active hepatitis or active liver disease other than NASH/NAFLD.
17. Alcoholic liver disease, as indicated by ANI > 0
18. Current use of anticoagulation therapy (such as warfarin) that cannot be discontinued for 7 days before and 14 days after the procedure.
19. Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 14 days before and 14 days after the procedure.
20. Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of acetaminophen and low dose aspirin is allowed.
21. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the baseline visit.
22. Use of drugs known to affect GI motility (e.g. Metoclopramide)
23. Use of weight loss medications such as Meridia, Xenical, Phentermine or over-the-counter weight loss medications (prescription medication)
24. Currently taking, or unable to stop taking dietary supplements or herbal agents, including vitamin C or multivitamins containing vitamin C at >500 mg per day, multivitamins containing biotin (vitamin B7), and supplements for hair, skin, and nail growth. Multivitamins not containing biotin are permitted.
25. Persistent anemia, defined as hemoglobin <10 g/dL.
26. Known history of hemoglobinopathy.
27. Known history of blood donation or transfusion within 3 months prior to the Screening Visit.
28. Known history of cardiac arrythmia
29. Significant cardiovascular disease, including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within 6 months prior to the Screening Visit.
30. Estimated glomerular filtration rate (eGFR) ≤ 60 ml/min/1.73m2 (estimated by MDRD).
31. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the participant a poor candidate for clinical trial participation in the opinion of the investigator.
32. History of secondary hypothyroidism or inadequately controlled primary hypothyroidism (TSH value outside the normal range at screening)
33. With any implanted electronic devices or duodenal metallic implants
34. Not a candidate for upper GI endoscopy or general anesthesia.
35. Active illicit substance abuse or alcoholism (>2 drinks/day regularly)
36. Active malignancy within the last 5 years (excluding non-melanoma skin cancers)
37. Women breastfeeding
38. Participating in another ongoing clinical trial of an investigational drug or device.
39. Any other mental or physical condition which, in the opinion of the study investigator, makes the participant a poor candidate for clinical trial participation.
40. Critically ill or has a life expectancy <3 years

    Additional exclusion criteria to be confirmed during the screening process:
41. HbA1c < 7.5% or > 10% at baseline visit
42. Any severe hypoglycemic event since the screening visit
43. CGM readings <54 mg/dl in more than 1% of time by CGM since the screening visit
44. CGM readings > 360 mg/dL in more than 1% of time
45. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic)
46. Women of child-bearing potential with a positive urine pregnancy test at baseline visit
47. LA Grade C or greater esophagitis on endoscopy
48. Abnormalities of the GI tract preventing endoscopic access to the duodenum
49. Anatomic abnormalities in the duodenum that would preclude the completion of the treatment procedure, including tortuous anatomy
50. Endoscopic observation of upper gastrointestinal abnormality such as ulcers, polyps, varices, strictures, congenital or intestinal telangiectasia
51. Any other anatomical or endoscopic abnormalities/characteristics that, in the opinion of the investigator, would preclude safe use of the investigational device or procedure

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2025-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DeMarco, MD, Study Chair — Baylor Scott & White
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - Cuyuna Regional Medical Center, Crosby, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 study sites in the US. Twenty participants were enrolled (i.e. received Endogenex treatment). Two participants did not complete the study due to patient withdrawal and physician withdrawal to relocation.
Pre-assignment Details: Pre-assignment did not occur in this study. All participants that met inclusion criteria and none of the exclusion criteria received treatment with the Endogenex device. At the time of the procedure, a screening endoscopy was performed on all participants to visually confirm the suitability of GI anatomy and excluding any participants with anatomy that met exclusion or preclude operator's ability to safely complete the treatment.
Groups:
- Interventional Arm- Endogenex (PEF) Treatment: Participants meeting inclusion and not meeting exclusion were treated with the Endogenex device. The Endogenex device is designed to induce duodenal mucosal regeneration using pulsed electric field via non-surgical, endoscopic approach.
Period: Overall Study
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Started | 20
Completed | 18 (2 participants were exited from the study at 24 weeks after completing the primary safety endpoint)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
Age, Customized [Mean (Standard Deviation); unit: years] — Mean Age (years)
  years
    Age | 54.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
HbA1c (%) [Mean (Standard Deviation); unit: %] | 8.3 (0.54)
Duration of Diabetes (years) [Mean (Standard Deviation); unit: years] | 6.7 (2)
BMI (kg/m²) [Mean (Standard Deviation); unit: kg/m²] | 32.4 (4.3)
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 224 (39)

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Device- or Procedure-Related Serious Adverse Events (SAE)
Description: Number of participants experiencing device- or procedure-related serious adverse events (SAE)
Time Frame: 12 weeks post-procedure
Population: Primary endpoint was performed at 12 weeks. At the 12 weeks, data from all 20 participants were available. Two participants exited the study at the 24 week visit, resulting in the 18 participants completing the study at 48 weeks.
Measure: Number; unit: Number of Participants with related SAE
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
Number of Participants with related SAE | 0

2. Secondary Outcome: Mean HbA1c by Follow-up Visit
Description: Mean HbA1c by Post Procedure Follow-up Visits
Time Frame: at 4,12, 24, and 48 Weeks Post Procedure
Population: Two participants were exited from the study by 24 weeks
Measure: Mean (Standard Deviation); unit: HbA1c %
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
HbA1c %
  Mean HbA1c at Week 4 Post Procedure | 7.2 (0.7)
  Mean HbA1c at Week 12 Post Procedure | 6.7 (0.7)
  Mean HbA1c at Week 24 Post Procedure: number analyzed (Participants) | 18
  Mean HbA1c at Week 24 Post Procedure | 6.9 (1.1)
  Mean HbA1c at Week 36 Post Procedure: number analyzed (Participants) | 18
  Mean HbA1c at Week 36 Post Procedure | 7.0 (0.7)
  Mean HbA1c at Week 48 Post Procedure: number analyzed (Participants) | 18
  Mean HbA1c at Week 48 Post Procedure | 7.2 (0.8)

3. Secondary Outcome: Mean Fasting Plasma Glucose (FPG) by Visit
Description: Mean Fasting Plasma Glucose (FPG) at Post Procedure Follow-up Visit
Time Frame: Follow-up at 4,12, 24, 36, and 48 weeks post procedure
Population: Two participants were exited from the study by 24 weeks.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
mg/dL
  Mean FPG at Week 4 post procedure | 140.1 (28.6)
  Mean FPG at Week 12 post procedure | 155.7 (28.8)
  Mean FPG at Week 24 post procedure: number analyzed (Participants) | 18
  Mean FPG at Week 24 post procedure | 155.9 (42.7)
  Mean FPG at Week 36 post procedure: number analyzed (Participants) | 18
  Mean FPG at Week 36 post procedure | 150.8 (24.2)
  Mean FPG at Week 48 at post procedure: number analyzed (Participants) | 18
  Mean FPG at Week 48 at post procedure | 161.6 (37.0)

4. Secondary Outcome: Mean Weight by Follow-up Visit
Description: Mean weight by Post Procedure Follow-up Visit
Time Frame: Follow-up at 4,12, 24, 36, and 48 weeks post procedure
Population: Two participants were exited by 24 Weeks
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
lbs
  Mean Weight at Week 4 Post Procedure | 215.6 (38.1)
  Mean Weight at Week 12 Post Procedure | 209.3 (36.1)
  Mean Weight at Week 24 Post Procedure: number analyzed (Participants) | 18
  Mean Weight at Week 24 Post Procedure | 214.9 (40.3)
  Mean Weight at Week 36 Post Procedure: number analyzed (Participants) | 18
  Mean Weight at Week 36 Post Procedure | 213.3 (41.1)
  Mean Weight at Week 48 Post Procedure: number analyzed (Participants) | 18
  Mean Weight at Week 48 Post Procedure | 217.8 (41.7)

5. Other Pre Specified Outcome: Procedural Success
Description: Percentage of participants with successful DMR procedure
Time Frame: At the time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
Participants | 20

6. Other Pre Specified Outcome: Procedural Time
Description: Time between catheter insertion to catheter removal
Time Frame: At the time of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
Number analyzed (Participants) | 20
minutes | 82.9 (20.1)

ADVERSE EVENTS:
Time Frame: Enrollment through study completion at 48 weeks
Arm/Group | Interventional Arm- Endogenex (PEF) Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm- Endogenex (PEF) Treatment (N=20)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) — Not device-related
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) — Not device-related
Cholecystectomy (Hepatobiliary disorders) | 1 (1) — Not device-related
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not device-related
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not device-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm- Endogenex (PEF) Treatment (N=20)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Upper abdominal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
CGM application site bleed (Skin and subcutaneous tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Conjunctivitis (Infections and infestations) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
COVID-19 (Infections and infestations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Vascular disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Hemmorrhoids (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Influenza like illness (Infections and infestations) | 1 (1)
Limb Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Lip Injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngititis (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Esophagititis (Gastrointestinal disorders) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1)
Oropharyngeal Pain (Gastrointestinal disorders) | 14 (14)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pharyngititis (Gastrointestinal disorders) | 1 (1)
Plantar Facititis (Musculoskeletal and connective tissue disorders) | 1 (1)
Polypectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Procedural Dizziness (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin Papilloma (Skin and subcutaneous tissue disorders) | 1 (1)
Toothache (General disorders) | 1 (1)
Ulcerative Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Lip Swelling (Injury, poisoning and procedural complications) | 1 (1)
Orthostatic Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This pilot study was designed to assesses the initial safety of the Endogenex device in participants with type 2 diabetes. Due to the small sample size, no formal hypothesis testing was performed. Descriptive statistics are reported using mean and standard deviations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT05014204/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05014204/SAP_001.pdf